CLINICAL TRIAL: NCT07348588
Title: Intravitreal Adalimumab in Inherited and Degenerative Retinal Diseases: A Prospective Comparative Pilot Study
Brief Title: Intravitreal Adalimumab in Inherited and Degenerative Retinal Diseases
Acronym: ADARET
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centro de Pesquisa Rubens Siqueira (Other)
Responsible Party: Principal Investigator, Rubens Camargo Siqueira, MD,PhD, Centro de Pesquisa Rubens Siqueira
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADARET
Record Dates: First submitted 2025-11-30; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Retinitis Pigmentosa (RP); Extensive Macular Atrophy With Pseudodrusen (EMAP)
Keywords: retinitis pigmentosa; intravitreal adalimumab; visual field; ERG; Ellipsoid zone; retinal degeneration
MeSH Terms: conditions — Retinitis Pigmentosa; Retinal Degeneration

STUDY DESIGN:
Intervention Model Description: his is a prospective, single-arm, open-label interventional pilot study designed to assess the ocular safety, feasibility, and functional outcomes of intravitreally administered adalimumab in patients with retinitis pigmentosa. All participants receive the same intervention-adalimumab 2 mg/0.05 mL-administered at baseline (M0), and at two-month intervals (M2, M4), for a total of three injections.
  Given the exploratory nature and rarity of the condition, no randomization or masking is applied. Each participant serves as their own control, with outcomes evaluated as within-subject pre-post changes from baseline to six months (M0-M6).
  The study is structured to provide proof-of-concept data regarding the therapeutic potential of local TNF-α inhibition in inherited retinal degenerations. This model prioritizes real-world applicability, tolerability, and early detection of functional trends (visual acuity, field sensitivity, ERG, and OCT biomarkers) to inform the design of future controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intravitreal injection of adalimumab (Experimental): Participants receive intravitreal injections of adalimumab 2 mg/0.05 mL at baseline (M0), month 2 (M2), and month 4 (M4).
  This arm evaluates the effect of anti-TNF-α immunomodulation alone on visual function and retinal structure in patients with Retinitis Pigmentosa and EMAP.
  Interventions: Drug: Intravitreal Adalimumab

INTERVENTIONS:
Drug: Intravitreal Adalimumab — Participants receive intravitreal injections of adalimumab 2 mg/0.05 mL at baseline (M0), month 2 (M2), and month 4 (M4).

SUMMARY:
This prospective, comparative pilot study investigates the safety and functional outcomes of intravitreal adalimumab (ADA) in patients with Retinitis Pigmentosa (RP) and Extensive Macular Atrophy with Pseudodrusen-like Appearance (EMAP).

Participants will receive three intravitreal injections of adalimumab (2 mg/0.05 mL) at two-month intervals (M0, M2, M4).

The primary objective is to assess functional changes after 6 months, focusing on visual-field preservation (Field Preservation Deviation Index - FPDI, Mean Deviation - MD) and best-corrected visual acuity (LogMAR).

Secondary outcomes include alterations in 30-Hz flicker ERG amplitude, OCT parameters (central macular thickness and ellipsoid zone length), and ocular safety measures such as intraocular pressure and inflammatory response.

DETAILED DESCRIPTION:
Retinitis pigmentosa (RP) represents a genetically and phenotypically heterogeneous group of inherited retinal dystrophies characterized by progressive photoreceptor degeneration, classically beginning with rod dysfunction and followed by cone loss. Patients typically present with nyctalopia, peripheral visual-field constriction, and, in advanced stages, central vision impairment. Despite significant advances in gene-specific, cell-based, and prosthetic approaches, most patients currently lack broadly applicable interventions capable of slowing or reversing disease progression across RP's wide genotypic spectrum.

Recent evidence reframes RP as not only a genetic degenerative process but also a state of chronic para-inflammation in the outer retina. Microglial activation, breakdown of the blood-retinal barrier, and overexpression of pro-inflammatory cytokines-particularly tumor necrosis factor-alpha (TNF-α)-have been implicated in accelerating photoreceptor apoptosis and secondary cone degeneration. Within this biological context, adalimumab (ADA), a fully human monoclonal antibody that selectively inhibits TNF-α, offers a mechanism-based therapeutic rationale for mitigating inflammatory injury in RP.

This prospective, single-arm pilot study was designed to evaluate the functional impact and ocular safety of intravitreal adalimumab in patients with RP. Participants received three intravitreal ADA injections (2 mg/0.05 mL) at two-month intervals (M0, M2, M4). The primary assessments included best-corrected visual acuity (BCVA, LogMAR), visual-field metrics (FPDI, MD, PSD; using 10-2 for advanced and 24-2 for less advanced disease), and 30-Hz flicker ERG when measurable. Structural endpoints comprised OCT-derived central macular thickness and ellipsoid zone (EZ) length. Outcomes were analyzed for pre-post change over six months (M0-M6) and feasibility in a real-world clinical research setting.

This exploratory study aims to generate foundational data to guide future controlled trials of anti-TNF therapy in inherited retinal degenerations with inflammatory components.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years.

* Clinical diagnosis of retinitis pigmentosa (RP) or EMAP (Extensive Macular Atrophy with Pseudodrusen-like Appearance) confirmed by multimodal evaluation.
* Best-corrected visual acuity (BCVA) ≥ counting fingers at 1 meter (approximately ≤ 1.9 logMAR) in the study eye.
* Measurable visual field on iCare COMPASS (10-2 or 24-2) with acceptable reliability indices.
* Clear ocular media adequate for safe intravitreal injection and high-quality OCT imaging.
* Ability and willingness to provide written informed consent.
* Ability to comply with scheduled study visits (Baseline [M0], Day 7-14 after injections, Month 2 [M2], Day 7-14, Month 4 [M4], Day 7-14, and Month 6 [M6]).
* For ERG subset only: presence of a recordable baseline 30-Hz flicker ERG response (signal-to-noise ratio ≥ 3:1 and amplitude ≥ 3.0 µV).
* Note: Absence of a measurable flicker ERG response does not exclude participation in the main study.

Exclusion Criteria:

* Active ocular inflammation (anterior, intermediate, or posterior uveitis) or infectious ocular disease in the study eye.
* Active choroidal neovascularization or other macular diseases unrelated to RP or EMAP.
* Uncontrolled glaucoma (intraocular pressure > 21 mmHg despite therapy) or optic neuropathies not related to RP or EMAP.
* Significant media opacity that may impair imaging quality or safe intravitreal injection.
* Recent ocular interventions that may confound study outcomes, including:
* Intravitreal therapy within 3 months prior to enrollment.
* Periocular corticosteroid injection within 3 months prior to enrollment.
* Major intraocular surgery within 3 months prior to enrollment.
* Known hypersensitivity to adalimumab, povidone-iodine, local anesthetics, or any formulation components.
* Coagulopathy or contraindications to ocular injections (platelet count < 100,000/µL or INR > 1.5 unless corrected).
* Pregnancy or breastfeeding.
* Women of childbearing potential unwilling to use effective contraception during the study period.
* Uncontrolled systemic disease that increases risk or interferes with study participation or completion.
* Participation in another interventional clinical trial within 3 months prior to enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Field Preservation Deviation Index (FPDI) | Baseline to Month 6
  Change (Δ) in Field Preservation Deviation Index (FPDI), expressed as a percentage (%), measured by automated perimetry using the iCare COMPASS system. The FPDI reflects the proportion of preserved visual field relative to age-matched normative data and provides a quantitative assessment of global visual field integrity. The outcome is defined as the difference between baseline (Month 0) and Month 6 values in the study eye.
Change in Mean Deviation (MD) | Baseline to Month 6
  Change (Δ) in Mean Deviation (MD), expressed in decibels (dB), measured by automated perimetry using the iCare COMPASS system. Mean Deviation represents the average difference in retinal sensitivity compared with age-adjusted normative values, serving as a global index of visual field loss. The outcome corresponds to the difference between baseline (Month 0) and Month 6 measurements in the study eye.
Change in Best-Corrected Visual Acuity (BCVA) | Baseline to Month 6
  Change (Δ) in Best-Corrected Visual Acuity (BCVA), expressed in logarithm of the minimum angle of resolution (LogMAR), measured using standardized Early Treatment Diabetic Retinopathy Study (ETDRS) charts under controlled testing conditions. BCVA assesses central visual function and foveal integrity. The outcome is defined as the difference between baseline (Month 0) and Month 6 BCVA values in the study eye.

SECONDARY OUTCOMES:
Change in Pattern Standard Deviation (PSD) | Baseline to Month 6
  Change (Δ) in Pattern Standard Deviation (PSD), expressed in decibels (dB), measured by automated perimetry using the iCare COMPASS system. PSD reflects localized irregularities in visual field sensitivity and is particularly sensitive to focal or non-uniform patterns of visual field loss. The outcome is defined as the difference between baseline (Month 0) and Month 6 measurements in the study eye.
Change in 30-Hz Flicker ERG Amplitude | Baseline to Month 6
  Change (Δ) in 30-Hz flicker electroretinogram (ERG) amplitude, expressed in microvolts (µV), measured in accordance with International Society for Clinical Electrophysiology of Vision (ISCEV) standards. The 30-Hz flicker ERG primarily assesses cone-mediated retinal function and provides an objective measure of global photoreceptor and post-receptoral pathway integrity. The outcome corresponds to the difference between baseline (Month 0) and Month 6 values in the study eye.
Change in Central Macular Thickness (CMT) | Baseline to Month 6
  Change (Δ) in central macular thickness (CMT), expressed in micrometers (µm), measured by spectral-domain optical coherence tomography (SD-OCT). CMT represents the average retinal thickness within the central macular subfield and serves as a structural biomarker of macular integrity, including retinal edema, atrophy, or remodeling. The outcome is defined as the difference between baseline (Month 0) and Month 6 measurements in the study eye.
Change in Ellipsoid Zone (EZ) Length | Baseline to Month 6
  Change (Δ) in ellipsoid zone (EZ) length, expressed in micrometers (µm), measured by spectral-domain optical coherence tomography (SD-OCT). EZ length reflects the integrity and spatial extent of photoreceptor inner segment ellipsoid band and is a sensitive structural biomarker of photoreceptor preservation in degenerative retinal diseases. The outcome corresponds to the difference between baseline (Month 0) and Month 6 measurements in the study eye.

CONTACTS AND LOCATIONS:
Locations (1):
- Rubens Siqueira Research Center, São José do Rio Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Siqueira RC, Brandao CC. The Role of Cytokines in Degenerative Retinal Diseases: A Comprehensive Review. Biomedicines. 2025 Jul 15;13(7):1724. doi: 10.3390/biomedicines13071724. PMID 40722794